CLINICAL TRIAL: NCT04085770
Title: Short Term Effect of Vitamin D Supplementation on the Clinical Outcomes in Patients Undergoing Valve Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sandra Nael Naguib Wahba, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CL(1686)
Record Dates: First submitted 2019-09-03; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Valve Replacement Complication
Keywords: LOS; mediastinitis; secondary myocardial infection
MeSH Terms: conditions — Mediastinitis | interventions — alfacalcidol

STUDY DESIGN:
Intervention Model Description: randomized ,controlled, open-label, parallel clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alfacalcidol (Experimental): Patients allocated to the alfacalcidol group received 2 mcg of oral Bone Care© soft gelatin capsules once daily with food starting from the day of admission till the end of hospital stay.
  Interventions: Drug: Alfacalcidol 1 MCG Oral Capsule
- Control (No Intervention): Control group were exposed to the same conditions as the treatment group except they were not given one-alfacalcidol.

INTERVENTIONS:
Drug: Alfacalcidol 1 MCG Oral Capsule — 2 mcg of oral Bone Care© soft gelatin capsules once daily with food starting from the day of admission till the end of hospital stay
  Other Names: Bone care
  Arms: Alfacalcidol

SUMMARY:
This study evaluates the effect of Vitamin D supplementation on ICU and hospital LOS in patients undergoing valve replacement surgery. Half of the patients will receive Alfacalcidol, while the other half-the control group- will be exposed to the same environment without receiving alfacalcidol.

DETAILED DESCRIPTION:
Vitamin D insufficiency has been reported in more than 80% of critically ill patients, hospitalized in intensive care unit (ICU), including cardiac surgical patients. Moreover, 25(OH)D levels continue to decrease from baseline throughout the hospital stay and resolves by 6 months. Vitamin D levels < 20 ng/ml is associated with higher mortality, infection rates and prolonged length of ICU saty.

The discovery of vitamin D receptors (VDR) expressed on cardiac muscle and vasculature, released a strong hypothesis suggesting that vitamin D regulates RAAS activity and cardiac remodeling.

The beneficial effects of vitamin D on cardiovascular system, immune function and wound healing could be of particular interest in critical care, and patients undergoing valve replacement surgery will benefit the most.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing mechanical valve replacement surgery

Exclusion Criteria:

* combined valvular replacement surgery and Coronary Artery Bypass Graft (CABG) surgery
* valvular replacement redo
* valvular replacement surgery secondary to infective endocarditis
* on dialysis
* ALT levels 2-3 times higher than normal range
* CHD,
* impaired gastrointestinal function
* indication for vitamin D supplementation within the prior month
* hypercalcemia defined as total calcium >10.4 mg/dl
* hyperphosphatemia defined as serum phosphate > 4.5 mg/dl
* pregnancy and lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
hospital length of stay | time to hospital discharge, up to 15 days
  length of hospital stay in days starting from ICU admission to hospital discharge.
intensive-care unite length of stay | time to ICU discharge, up to 7 days
  length of hospital stay in hours starting from ICU admission to ICU discharge.

SECONDARY OUTCOMES:
Rate of postoperative complications | during hospital stay, up to 15 days
  compare rate of postoperative infections, decline in LV functions, MI or massive bleeding between the 2 arms
mortality | during hospital stay, up to 15 days
  compare mortality rate between the 2 arms
monitor alfacalcidol safety | during hospital stay, up tp 15 days
  the measurement of alfacalcidol blood concentration indirectly through the measurement of serum 25(OH)D and monitoring of its metabolic effect through the measurement of serum total calcium and phosphorous

CONTACTS AND LOCATIONS:
Locations (1):
- El-Demerdash Cardiac Academy Hospital, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naguib SN, Sabry NA, Farid SF, Alansary AM. Short-term Effects of Alfacalcidol on Hospital Length of Stay in Patients Undergoing Valve Replacement Surgery: A Randomized Clinical Trial. Clin Ther. 2021 Jan;43(1):e1-e18. doi: 10.1016/j.clinthera.2020.11.008. Epub 2020 Dec 16. PMID 33339609